CLINICAL TRIAL: NCT01426828
Title: Randomized Phase II Trial of CD3/CD28 Activated Id-KLH Primed Autologous Lymphocytes in Subjects With Myeloma Undergoing Autologous Transplant
Brief Title: Id-KLH Vaccine + T Cells in Subjects With Myeloma Undergoing Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 07409
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Results first posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Multiple Myeloma
Keywords: adult; symptomatic multiple myeloma; myeloma; diagnosis within 12 months of initiation of systemic therapy
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Other): Arm A will receive the CD3/CD28 activated autologous lymphocytes intravenously and subcutaneous injections of "KLH only" vaccine.
  Interventions: Biological: CD3/CD28
- Arm B (Other): Arm B will receive the CD3/CD28 activated autologous lymphocytes intravenously and subcutaneous injections of ID-KLH Vaccine Myeloma Immunoglobulin Idiotype Vaccine (id-KLH vaccine)
  Interventions: Biological: CD3/CD28

INTERVENTIONS:
Biological: CD3/CD28 — CD3/CD28 activated autologous lymphocytes intravenously

SUMMARY:
This study will enroll myeloma subjects undergoing autotransplantation. The primary objective of this study is to evaluate whether infusions of Id-KLH primed CD3/CD28 activated autologous lymphocytes mediate a more intense Id-specific immunity than non Id-KLH primed CD3/CD28 activated autologous lymphocytes. There will be 2 arms in the study, one receiving a DLI with non Id-KLH vaccine and one receiving aDLI with Id-KLH vaccine.

DETAILED DESCRIPTION:
The primary objectives of this study is to evaluate whether infusions of Id-KLH primed CD3/CD28 activated autologous lymphocytes mediate a more intense id-specific immunity than non id-KLH primed CD3/CD28 activated autologous lymphocytes. The secondary objectives of this study is to demonstrate that doses of 1 times 10e10 Id-KLH primed CD3/CD28 autologous lymphocytes can be infused safely and effectively in more than 80 percent of eligible patients, to determine whether Id-KLH primed CD3/CD28 activated autologous lymphocytes and to determine if the presence of Id-specific immunity correlates with disease response.

ELIGIBILITY:
Inclusion Criteria:

SCREEN #1 (Visit 1) Step 1:

* Diagnosis of symptomatic multiple myeloma.
* Less than 10 months after initiation of systemic therapy.
* One or two lines of induction therapy with commonly used regimens.
* Age greater than or equal to 18 years to less than or equal to 70 years at the time of enrollment.
* IgG paraprotein (not of IgG3 subtype) with a paraprotein peak (M-spike) of ≥0.2 g/dL. Alternatively subjects who have previously stored purified Id-specific protein on other clinical or laboratory protocols.
* Echocardiogram or MUGA with an ejection fraction of 45% or more and no uncompensated congestive heart failure or uncontrolled arrhythmias.
* Adequate pulmonary function as defined by FEV1, FVC and actual or corrected DLCO of 50% or greater of the predicted value for age, sex and size.
* Adequate renal function as defined by creatinine of 2.0 mg/dl or less or a creatinine clearance of 40cc/min or more.
* Adequate hepatic function as defined by a total bilirubin of 2.0 mg/dl or less and AST and ALT less than 2 times upper limit of normal.
* Ability to sign written informed consent.
* Karnofsky performance status of at least 80% or more.
* Negative serum Beta HCG test in women of child bearing potential and agree to use a medically acceptable form of birth control while on the study drugs.

Exclusion:

* Subjects with melphalan-based induction
* Active uncontrolled infection
* HIV+ or active hepatitis B or C as defined by positive viral load or serology.
* Pre-existing autoimmune diseases, with exception of Hashimoto's thyroiditis.
* Concurrent use of systemic steroids at the time of cell infusion or cell collection, or a condition, in the treating physician's opinion, that is likely to require steroid therapy during Tcell collection or after infusion. Steroids for disease treatment at times other than cell collection or at the time of infusion are permitted. Use of inhaled steroids is permitted as well.
* Prior autologous or allogeneic transplant.

For this study, there will be no exceptions to eligibility granted.

4.2 PRE-VACCINE #1 ASSESSMENT (Visit 3) Step 2

Subjects must meet the following criteria to proceed with vaccination:

* Less than 9 months from randomization.
* Adequate renal function as defined by creatinine of 2.0 mg/dl or less or a creatinine clearance of 40cc/min or more.
* Adequate hepatic function as defined by a total bilirubin of 2.0 mg/dl or less and AST and ALT less than 2 times upper limit of normal.
* Karnofsky performance status of at least 80% or more.
* At least 2 weeks from last chemotherapy.
* Negative serum Beta HCG test in women of child bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2016-06 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ed Stadtmauer, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine; Muzaffar H. Qazilbash, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas, MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Qazilbash MH, Saini NY, Cha SC, Wang Z, Stadtmauer EA, Baladandayuthapani V, Lin H, Tross B, Honhar M, Rao SS, Kim K, Popescu M, Szymura S, Zhang T, Anderson A, Bashir Q, Shpall EJ, Orlowski RZ, Levine BL, Kerr N, Garfall A, Cohen A, Vogl DT, Dengel K, June CH, Champlin R, Kwak LW. A randomized phase 2 trial of idiotype vaccination and adoptive autologous T-cell transfer in patients with multiple myeloma. Blood. 2022 Mar 3;139(9):1289-1301. doi: 10.1182/blood.2020008493. PMID 34521108

RESULTS

PARTICIPANT FLOW:
Period: Overall Study Evaluations
Arm/Group | Arm A | Arm B
Started | 22 | 18
Completed | 17 | 15
Not Completed | 5 | 3
Period: Immune Response Analysis
Arm/Group | Arm A | Arm B
Started | 17 | 15
Completed (Only those subjects that had sufficient PBMC samples from pre-vaccination (D0), and Day 30, Day 90 and Day 180 time points for NanoString gene expression analysis were included in the immune response analysis.) | 8 | 8
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 13 | 29
  >=65 years | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 13 | 10 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 19 | 14 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Participants With Id-specific Immunity
Description: Evaluate whether infusions of Id-KLH primed CD3/CD28 activated autologous lymphocytes mediate a more intense Id-specific immunity than non Id-KLH primed CD3/CD28 activated autologous lymphocytes. RNA was isolated from CD4 and CD8 T cells pre-vaccine, and at day 30, 90 and 180 post-vaccine for gene expression analysis. The Nanostring Human immunology V2 kit, a multiplex assay for 594 genes involved in the human immunology response, was used with an nCounter digital analyzer to quantify immune response gene expression levels. Subjects were considered to have Id-specific immunity if they induced expression of effector (TBX21, KLRG1) and memory (CCL5) associated genes in CD8 T cells in post-vaccine time-points compared to baseline.
Time Frame: 180 DAYS
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 8 | 8
Participants | 0 | 8

ADVERSE EVENTS:
Time Frame: 1 year
Description: The adverse event data included below reflects all data that can currently be verified by the sponsor. There is additional data that has yet to be verified by the investigator that will be included when available.
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18
Serious Adverse Events (participants affected / at risk) | 6/22 | 4/18
Other Adverse Events (participants affected / at risk) | 20/22 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=22) | Arm B (N=18)
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Fever (General disorders) | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Infections and infestations - Other (Influenza A) (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Skin and subcutaneous tissue disorders - Other (Sweet's syndrome) (Skin and subcutaneous tissue disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=22) | Arm B (N=18)
Anemia (Blood and lymphatic system disorders) | 11 | 7
Anorexia (Metabolism and nutrition disorders) | 2 | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Chills (General disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Diarrhea (Gastrointestinal disorders) | 11 | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Edema limbs (Gastrointestinal disorders) | 5 | 0
Fatigue (Gastrointestinal disorders) | 11 | 10
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 2
Fever (General disorders) | 6 | 6
General disorders and administration site conditions - Other (Achiness at injection site) (General disorders) | 2 | 0
General disorders and administration site conditions - Other (Body aches) (General disorders) | 2 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 | 3
Headache (Nervous system disorders) | 4 | 5
Hypokalemia (Metabolism and nutrition disorders) | 2 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 2
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 0
Hypotension (Vascular disorders) | 2 | 2
Infections and infestations - Other (C.Diff) (Infections and infestations) | 2 | 0
Injection site reaction (General disorders) | 6 | 4
Insomnia (Psychiatric disorders) | 5 | 2
Lymphocyte count decreased (Investigations) | 6 | 3
Mucositis oral (Gastrointestinal disorders) | 6 | 6
Nausea (Gastrointestinal disorders) | 15 | 12
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Neutrophil count decreased (Investigations) | 8 | 6
Oral pain (Gastrointestinal disorders) | 2 | 0
Pain (General disorders) | 5 | 0
Papulopustular rash (Infections and infestations) | 3 | 4
Platelet count decreased (Investigations) | 12 | 10
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper respiratory infection (Infections and infestations) | 2 | 0
Vomiting (Gastrointestinal disorders) | 7 | 8
Weight gain (Investigations) | 2 | 0
White blood cell decreased (Investigations) | 13 | 7
Alanine aminotransferase increased (Investigations) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Blood bilirubin increased (Investigations) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 2
Esophagitis (Gastrointestinal disorders) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
Unable to obtain finalized adverse event information from external site. Adverse event information is from the Annual Report submitted to the FDA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No